CLINICAL TRIAL: NCT06803732
Title: Postoperative Pain of Robotic, Endoscopic and Open Lateral Neck Dissection
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Zhan, Principal Investigator, Shanghai 6th People's Hospital
Other Study IDs: 2025-KY-095(K)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative; Thyroid Diseases; Surgery
Keywords: Lateral neck dissection; Robotic thyroid surgery; Minimally invasive surgery
MeSH Terms: conditions — Pain, Postoperative; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic group: Patients underwent lateral neck dissection via robotic approach
  Interventions: Other: Observations on postoperative pain intensity
- Endoscopic group: Patients underwent lateral neck dissection via endoscopic approach
  Interventions: Other: Observations on postoperative pain intensity
- Open group: Patients underwent lateral neck dissection via open approach
  Interventions: Other: Observations on postoperative pain intensity

INTERVENTIONS:
Other: Observations on postoperative pain intensity — pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain on operation day, postoperative day 1, postoperative month 1, postoperative month 3

SUMMARY:
Postoperative pain is a good indicator to confirm the advantages of the surgical methods in the era of minimally invasive surgery. Lateral neck dissection requires extensive dissection which may leads to postoperative numbness and pain. Robotic thyroid surgery has the advantage of precise and careful dissection and avoid the L-shape incision in the open approach. The study aims to explore the pain intensity and severity of lateral neck dissection on operation day, postoperative month 1 and postoperative month 3 among the robotic, endoscopic and open approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent lateral neck dissection via robotic, endoscopic or open approach
* Clinical diagnosis of differentiated thyroid cancer
* Clinical diagnosis of metastatic lateral lymph nodes

Exclusion Criteria:

* Participants with distant metastasis
* Participants with history of neck surgery or radiation
* Participants with vocal fold fixation by preoperative fibrolaryngoscope

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FNA proven differentiated thyroid cancer and metastatic lateral lymph nodes, underwent lateral neck dissection via robotic, endoscopic or open approach. Patients were well informed about the potential benefits and risks of robotic, endoscopic and open approach. Patient consented for us to use perioperative data.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
degree of pain | approximately 4 hours after surgery, on postoperative day 1, postoperative month 1 and postoperative month 3
  pain intensity was assessed using a standard visual analogue score, with a score of 0 to 10 corresponding to no pain to the most severe pain
Number of participants with recurrent laryngeal nerve injury | through study completion, an average of 1 year
  impaired vocal cord mobility confirmed by postoperative laryngoscopy
Number of participants with hypoparathyroidism | through study completion, an average of 1 year
  a postoperative parathyroid hormone level of less than 10 pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ling Zhan, Dr, Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request due to privacy or other restrictions. The data that support the findings of this study are available on request from Ling Zhan. The data are not publicly available due to them containing information that could compromise research participant privacy.